CLINICAL TRIAL: NCT03106831
Title: Small Doses of Pituitrin Versus Norepinephrine for the Management of Vasoplegic Syndrome in Patients After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Director of Center for Cardiac Intensive Care, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PX2016007
Record Dates: First submitted 2017-03-31; First posted 2017-04-10 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Postoperative Vasoplegic Syndrome
MeSH Terms: conditions — Vasoplegia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pituitrin arm (Experimental): To begin with 0.02 U/min to maintain mean arterial pressure(MAP) higher than 65 mmHg.
  Interventions: Drug: Pituitrin infusion
- Norepinephrine arm (Experimental): To begin with 0.04 μg/kg.min to maintain mean arterial pressure(MAP) higher than 65 mmHg.
  Interventions: Drug: Norepinephrine infusion

INTERVENTIONS:
Drug: Pituitrin infusion — To begin with 0.02 U/min to maintain mean arterial pressure(MAP) higher than 65 mmHg.
  Arms: Pituitrin arm
Drug: Norepinephrine infusion — To begin with 0.04 μg/kg.min to maintain mean arterial pressure(MAP) higher than 65 mmHg.
  Arms: Norepinephrine arm

SUMMARY:
Vasoplegic syndrome is a common complication after cardiac surgery. Low dose vasopressin can up-regulate blood pressure and improve clinical outcomes compared with norepinephrine (mainly acute kidney injury Anesthesiology 2017; 126:85-93). Pituitrin is used as a substitute for vasopressin in our center, which contains both vasopressin and oxytocin. Oxytocin may alleviate inflammatory process-associated kidney injury (Peptides 2006;27:2249-57). Therefore, the investigators hypothesize Pituitrin may be preferable to norepinephrine in the renal protection of patients with vasoplegic syndrome after cardiac surgery. Moreover, the serum levels of vasopressin, catecholamine, corticosteroid and corticotropin-releasing hormone will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as vasoplegic syndrome(defined as mean arterial pressure less than 65 mmHg resistant to fluid challenge and cardiac index greater than 2.2 L/min · m2) within 24 hours after cardiac surgery.

Exclusion Criteria:

1. Age < 18 and > 75 years.
2. Received renal replacement therapy before cardiac surgery.
3. Diagnosed as endocrine disease before cardiac surgery.
4. Diagnosed as sever peripheral vascular disease before cardiac surgery.
5. Extracorporeal membrane oxygenation support before admission.
6. To receive heart transplantation.
7. Infection on admission.
8. Pregnant or maternal patients.
9. Refusal of consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of in-hospital acute renal injury | 30 days
  Acute renal injury (AKI) is defined as any of the following: (1) increase in serum creatinine (SCr) by ≥ 26.5lmol/l in 48 hours; (2) increase in SCr to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or (3) urine output < 0.5 ml/kg/h for 6 hours (urine output is only assessed when the CRRT machine is absent or with a fluid removal rate of 0 ml/h).

SECONDARY OUTCOMES:
In-hospital mortality | 30 days
  All-cause mortality
Rate of new arrhythmias | 30 days
  Rate of new arrhythmias after cardiac surgery
Hormone levels | 30 days
  Serum hormone levels after cardiac surgery, including vasopressin, catecholamine, corticosteroid and corticotropin-releasing hormone
Rate of ECMO or LVAD support | 30 days
  Receiving extracorporeal membrane oxygenation (ECMO) or left ventricle assist device (LVAD) support
Duration on ventilator support | 30 days
  Duration on ventilator support after cardiac surgery
ICU length of stay | 30 days
  ICU length of stay
Hospital length of stay after cardiac surgery | 30 days
  Hospital length of stay after cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cardiac Intensive Care, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No